CLINICAL TRIAL: NCT05143814
Title: A Prospective Cohort Study Investigating the Success Rate of Fit Testing Following the Use of a 3D Printed Respirator Adapter From a Facial 3D Scan.
Brief Title: 3D Printed Mask Adapter Designed From Facial 3D Scans for Fit Testing.
Status: Withdrawn | Type: Observational
Why Stopped: COVID-19 suspension non-urgent studies
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 289974
Record Dates: First submitted 2021-11-23; First posted 2021-12-03 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: 3D Printed Mask Adapter Designed from Facial 3D scans for Fit testing. — Given the high level of fit test failures, without the provision of improved fits of masks, patient care will be highly curtailed for frontline staff at risk of SARS-CoV-2. Therefore, a reusable bespoke mask adapter used with a soft FFP3 disposable mask might be an economical solution to address the passing of fit testing. Currently, this is a major challenge in delivery of healthcare and urgent action is needed.

SUMMARY:
Healthcare workers PPE (personal protective equipment) when interacting with patients either infected or, potentially carrying SARS-CoV-2. One of the major routes of transmission is via droplet spread through oral and nasal mucosa therefore respiratory protective equipment (RPE) is an important part of PPE. There are concerns in dentistry that droplet spread can be increased during aerosol-generating procedures (AGP). This poses an increased risk to dentists and allied professionals in a clinical setting.

Fit testing is needed to ensure a mask forms a facial seal around the mouth and nose. Using a respirator mask without fit testing can reduce its effectiveness from between 6-88% with an optimal facial seal being more critical than the filtering performance. Commercial respirator masks are mass-produced for ' standard' faces, and often fail to provide a good fit for users thereby compromising the intended respirator filtering capability.

Given the high level of fit test failures, without the provision of improved fits of masks, patient care will be highly curtailed for frontline staff at risk of SARS-CoV-2. Therefore, a reusable bespoke 3D printed mask adapter used with a soft FFP3 disposable mask provides an economical solution to address the passing of fit testing.

Barts Health NHS Trust staff members who have previously failed the fit test to the first line FFP3 disposable respirator will be invited to enrol in this study.

Barts/QMUL scan App will be used to capture the facial scan of the subjects using a research allocated smartphone. Participants will be asked to be clean-shaven without any facial jewellery which could hinder the scan data. The App automatically generates a customized 3D print file (.stl) which will be sent for 3D printing.

The mask adapter will be fitted over the first-line FFP3 respirator once it is properly worn and checked as per the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who would have previously failed the quantitative fit test on the Trust's first line FFP3 disposable respirator.
* Subjects willing to use a flexible, disposable FFP3 mask.
* Subjects should be a minimum of 18 years old.

Exclusion Criteria:

* Subjects unwilling or unable to give written consent.
* Subjects who cannot remove their facial hair for religious or other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare staff in Barts Healthy NHS trust who meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-02-25 (Estimated)

PRIMARY OUTCOMES:
The success of of fit testing will be measured and reported quantitively using a TSI portacount | 20 minutes mask fit test

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, London, United Kingdom